CLINICAL TRIAL: NCT06721078
Title: Evaluation of Long-Acting Injectable (LAI) and Teen Clubs in Adolescents (ATTUNE).
Acronym: ATTUNE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Africa Health Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A0005-6490/2023; 1UG1MD019435-01 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Hiv
Keywords: peer navigation; long acting injectables; antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: In Stage 1, we will evaluate the peer navigation intervention in a stepped-wedge, cluster-randomised trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer navigation effectiveness (Other): To determine the effectiveness of peer navigation on viral suppression and retention in care among adolescents living with HIV in South Africa.
  Interventions: Behavioral: Peer navigation effectiveness

INTERVENTIONS:
Behavioral: Peer navigation effectiveness — To determine the effectiveness of peer navigation on viral suppression and retention in care among adolescents living with HIV in South Africa.

SUMMARY:
This is a 2-stage study assessing the effect of peer navigation (support from peers) and long-acting injectable antiretroviral therapy (ART) on viral suppression and retention in care among adolescents living with HIV and receiving care in South Africa.

DETAILED DESCRIPTION:
This study aims to deploy peer-navigated support (psychosocial support, HIV education, appointment reminders, adherence support, sexual and reproductive health, and healthcare navigation) to facilitate viral suppression and retention in care as adolescents living with HIV transition into adult care. The study population includes adolescents from South Africa aged 12 to less than 19 years, living with HIV, aware of their HIV status and receiving ART for at least six months.

In Stage 1, the peer navigation intervention in a stepped-wedge, cluster-randomised trial implemented over 18 months in three 6-month steps across 12 clinics will be evaluated. In addition, during Stage 1, user and key stakeholder preferences will be evaluated for the uptake and use of long-acting injectable ART, perform a costing and economic analysis and a program evaluation of the public health impact of the intervention. In Stage 2, an individually-randomised trial will be nested in a subset of clinics to evaluate long-acting injectable ART in adolescents with HIV.

The study procedures include a peer navigation intervention in Stage 1, alongside a user and key stakeholder preferences evaluation for the uptake and use of long-acting injectable ART and a cost and economic evaluation.

The study duration is three years (about 7 visits). The stepped-wedge trial will be implemented in the first 18 months, after which participants will be followed for an additional 18 months to assess the sustainability of the intervention. The nested individually-randomised trial of long-acting ART will be conducted during the second 18-month period.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 - 19, at enrolment
* Living with HIV
* Aware of their HIV status
* Receiving ART for at least six months
* Able to read and/or speak English, isiZulu, Sepedi, Afrikaans, Xhosa, or Sesotho
* Willing and able to consent to study activities
* Willing and able to get parental consent for study activities
* (Stage 1, objective 2 only) Age ≥ 18 years and Caregiver of an adolescent with HIV
* (Stage 1, objective 2 only) Age ≥ 18 years and provides clinical services or is a policy maker involved in adolescents with HIV

Exclusion Criteria:

* Inability to read and/or speak English, isiZulu, Sepedi, Afrikaans, Xhosa, or Sesotho
* Severe mental or physical illness preventing participation in informed consent activities.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Peer navigation - viral suppression (effectiveness) | 18 months
  To determine the effectiveness of peer navigation on viral suppression among adolescents living with HIV in South Africa using the endpoint of viral load suppression (VL <50 copies/ml) over 18 months.
Peer navigation - retention in care (effectiveness) | 18 months
  To determine the effectiveness of peer navigation on retention among adolescents living with HIV in South Africa using the endpoint of retention (at least 1 health care visit in the last 90 days) over 18 months.

SECONDARY OUTCOMES:
Peer navigation - viral suppression (sustainability) | 36 months
  To assess the sustainability of the impact of peer navigation on viral suppression among adolescents living with HIV in South Africa using the endpoint of viral load suppression (VL <50 copies/ml) at 24 months and 36 months.
Peer navigation - retention (sustainability) | 36 months
  To assess the sustainability of the impact of peer navigation on retention in care among adolescents living with HIV in South Africa using the endpoint of retention (at least 1 health care visit in the last 90 days) at 24 months and 36 months.
long-acting injectable ART - acceptability | 36 months
  To identify the preferred user characteristics influencing the acceptability of long-acting injectable ART for adolescents with HIV with a qualitative evaluation of preferred user characteristics. Nine focus group discussions (FGDs) will be conducted with key stakeholders (caregivers of ALHIV, ALHIV ages 12 to less than 19, and adolescent HCWs/policy makers) to identify preferred user characteristics.
Economic evaluation analysis of providing LAI | 36 months
  The cost analysis and economic impact of long-acting injectable antiretroviral therapy on viral suppression and care retention in adolescents living with HIV and receiving care in South Africa. Average per patient treated per year; average cost per patient retained; average cost per patient virally suppressed; incremental cost per additional person virally suppressed; incremental cost per additional person retained; incremental cost per life year saved (ART)
Economic evaluation analysis of providing peer navigation | 36 months
  The cost analysis and economic impact of peer navigation on viral suppression and care retention in adolescents living with HIV and receiving care in South Africa. Average per patient treated per year; average cost per patient retained; average cost per patient virally suppressed; incremental cost per additional person virally suppressed; incremental cost per additional person retained; incremental cost per life year saved (ART).
Cost-effectiveness analyses of providing LAI | 36 months
  A time and motion evaluation will be conducted. The estimated average staff time-spend with patients triangulated with the cost of clinical staff salaries from public sector salaries, the type and number of laboratory tests per patient (patient medical records), and cost per test (National Health Laboratory Service, NHLS). Medication costs will also be monitored (patient medical records, published national drug unit costs), and consumable resources will be used during study procedures (staff interviews, government tenders from the National Department of Health, National Treasury). The total floor space required for the study will be calculated, and a market-related average rental cost per square meter will be applied to estimate the cost of the building. Utility costs will be obtained for the facility and applied by square meter.
Cost-effectiveness analyses of providing peer navigation | 36 months
  A time and motion evaluation will be conducted. The estimated average staff time-spend with patients triangulated with the cost of clinical staff salaries from public sector salaries, the type and number of laboratory tests per patient (patient medical records), and cost per test (National Health Laboratory Service, NHLS). Medication costs will also be monitored (patient medical records, published national drug unit costs), and consumable resources will be used during study procedures (staff interviews, government tenders from the National Department of Health, National Treasury). The total floor space required for the study will be calculated, and a market-related average rental cost per square meter will be applied to estimate the cost of the building. Utility costs will be obtained for the facility and applied by square meter.

OTHER OUTCOMES:
Providing long-acting injectable ART and peer navigators | 36 months
  Using the RE-AIM framework, determine the implementation factors involved in providing peer navigation and long-acting injectable ART during adolescent-friendly clinics across multiple settings in South Africa. Based on the implementation science framework RE-AIM, the Reach (enrolment in each region), Effectiveness (viral suppression and retention in care), Adoption (uptake at each regional clinic, acceptability, and feasibility), Implementation (fidelity to protocol) and Maintenance (sustainability and costing) of the interventions will be measured using the implementation strategies of peer navigation and audit and feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Moherndran Archary, PhD, Principal Investigator — Africa Health Research Institute